CLINICAL TRIAL: NCT04544124
Title: Expanding Capacity in Alberta to Deliver Contingency Patient Management in Outpatient Addiction Treatment: A Randomized Clinical Trial for Methamphetamine Use
Brief Title: Delivering Contingency Management in Outpatient Addiction Treatment
Acronym: PRISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, David Hodgins, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200443; 2021-HQ-000013 (Other Grant/Funding Number: Health Canada)
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Methamphetamine; Methamphetamine Abuse; Methamphetamine-dependence; Contingency Management; Substance Use; Substance Abuse; Substance Use Disorders; Drug Use; Drug Abuse; Adults; Humans
Keywords: Contingency Management; Methamphetamine; Substance Use; Treatment; Internet-Based Intervention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants who use methamphetamine and participants who use substances other than methamphetamine will randomly be assigned to one of two treatment arms: contingency management which incentivizes participants for their treatment attendance or treatment-as-usual with no contingency management.
Masking Description: Given incentivization will occur for attendance, it is not possible to blind conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency management for treatment attendance (Experimental): Participants who receive contingency management in addition to their usual care (treatment-as-usual). These participants are in the 12-week contingency management program which provides incentives for their treatment attendance.
  Interventions: Behavioral: Contingency management
- Treatment-as-usual (No Intervention): Participants who solely receive their usual care (treatment-as-usual) and do not receive contingency management.

INTERVENTIONS:
Behavioral: Contingency management — Incentives will be provided for treatment attendance over a 12-week period.
  Arms: Contingency management for treatment attendance

SUMMARY:
Methamphetamine misuse has become a growing concern in Alberta, creating a burden on the health care system. Further, individuals who use methamphetamine in Alberta exhibit significant difficulty remaining in treatment. These troubling patterns necessitate the provision of evidence-based practices (EBPs)-those grounded in empirical evidence-to ensure the best possible care and outcomes for those struggling with this addiction. Within the field of substance use (SU), contingency management (CM) is an extensively studied evidence-based treatment (EBT) for addictive disorders.

CM is an intervention that provides incentives to encourage positive behavioural change. Compared to standard care (treatment-as-usual (TAU)), CM has resulted in improvements in abstinence, attendance, adherence, retention, and quality of life. The efficacy of CM has largely been investigated in the context of reinforcing abstinence, though the literature suggests that CM which reinforces attendance may be as effective. Research from the US has examined the cost-effectiveness of CM and found that although CM costs more, it was associated with greater abstinence, treatment completion, and substance-absent urine compared to TAU. Despite the promising literature, the uptake of CM in Canada is limited making it difficult to understand whether this EBT is equally efficacious as compared to the US.

This study will implement and evaluate the efficacy of virtually delivered attendance-based CM in outpatient addiction treatment in Alberta. Participants (N=544) will be individuals seeking treatment for methamphetamine use (n=304) and individuals seeking treatment for substance use issues other than methamphetamine use (n=240). It is hypothesized that compared to participants in TAU, participants in CM will evidence: (1) greater retention, (2) greater attendance, (3) greater abstinence from methamphetamine and less methamphetamine use, (4) greater abstinence from other SU and less SU, and (5) greater improvement in quality of life over the intervention and follow-up periods. Exploratory aims include understanding how: outcomes differ based remote versus in-person delivery of CM; outcomes differ between participants who use methamphetamine and participants who use substances other than methamphetamine; the costs of CM differ from TAU; CM changes health service use.

ELIGIBILITY:
Inclusion Criteria:

* 18-years of age or older
* Seeking treatment for methamphetamine use or substance use issues other than methamphetamine use
* Reported methamphetamine use or substance use other than methamphetamine use within 3-months prior to study entry
* Deemed appropriate for treatment-as-usual using Alberta Health Services clinical procedures
* Willing to participate in the 12-week intervention in-person or virtually at least once weekly
* Willing to participate in-person or virtually for a follow-up at 3, 6, and 12-months following the 12-week intervention period
* Willing to complete questionnaires weekly during the 12-week intervention period and at each follow-up at 3, 6, and 12-months following the 12-week intervention period

Exclusion Criteria:

* Past or current history of gambling problems
* Imminent plans to enter an environment in which participation in this study is restricted (e.g., residential treatment, inpatient unit, detoxification, incarceration, house arrest).
* Attended more than one treatment session since their intake, or screening date was more than one month following their first day of treatment at the Alberta Health Services clinic
* No plans to attend weekly treatment at the Alberta Health Services clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Differences in Treatment Retention from Baseline to Post-Intervention at Week 12 | Baseline to Post-Intervention at Week 12.
  The number of days between the first and last scheduled treatment session.

SECONDARY OUTCOMES:
Proportion of Methamphetamine Abstinent Days Measured Using the Timeline Followback (TLFB) Questionnaire | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The TLFB is an instrument that assesses retrospective substance use. Abstinence from and use of methamphetamine will be examined using the TLFB based on Robinson and colleagues' definitions (2014) over the intervention period and follow-up periods.
Longest Consecutive Days of Methamphetamine Abstinence Measured Using the Timeline Followback (TLFB) Questionnaire | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The TLFB is an instrument that assesses retrospective substance use. Abstinence from and use of methamphetamine will be examined using the TLFB based on Robinson and colleagues' definitions (2014) over the intervention period and follow-up periods.
Longest Consecutive Days of Methamphetamine Use Measured Using the Timeline Followback (TLFB) Questionnaire | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The TLFB is an instrument that assesses retrospective substance use. Abstinence from and use of methamphetamine will be examined using the TLFB based on Robinson and colleagues' definitions (2014) over the intervention period and follow-up periods.
Proportion of Days Abstinent from Other Licit and Illicit Substances Measured Using the Timeline Followback (TLFB) Questionnaire | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The TLFB is an instrument that assesses retrospective substance use. Abstinence from and use of other licit and illicit substances will be examined using the TLFB based on Robinson and colleagues' definitions (2014) over the intervention period and follow-up periods.
Longest Consecutive Days Abstinent from Other Licit and Illicit Substances Measured Using the Timeline Followback (TLFB) Questionnaire | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The TLFB is an instrument that assesses retrospective substance use. Abstinence from and use of other licit and illicit substances will be examined using the TLFB based on Robinson and colleagues' definitions (2014) over the intervention period and follow-up periods.
Longest Consecutive Days of Use of Other Licit and Illicit Substances Measured Using the Timeline Followback (TLFB) Questionnaire | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The TLFB is an instrument that assesses retrospective substance use. Abstinence from and use of other licit and illicit substances will be examined using the TLFB based on Robinson and colleagues' definitions (2014) over the intervention period and follow-up periods.
Mean Number of Units Consumed of Other Quantifiable Licit and Illicit Substances Measured Using the Timeline Followback (TLFB) Questionnaire | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The TLFB is an instrument that assesses retrospective substance use. Abstinence from and use of other licit and illicit substances will be examined using the TLFB based on Robinson and colleagues' definitions (2014) over the intervention period and follow-up periods.
Total Number of Units Consumed of Other Quantifiable Licit and Illicit Substances Measured Using the Timeline Followback (TLFB) Questionnaire | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The TLFB is an instrument that assesses retrospective substance use. Abstinence from and use of other licit and illicit substances will be examined using the TLFB based on Robinson and colleagues' definitions (2014) over the intervention period and follow-up periods.
Largest Number of Units Consumed of Other Quantifiable Licit and Illicit Substances in One Day Measured Using the Timeline Followback (TLFB) Questionnaire | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The TLFB is an instrument that assesses retrospective substance use. Abstinence from and use of other licit and illicit substances will be examined using the TLFB based on Robinson and colleagues' definitions (2014) over the intervention period and follow-up periods.
Proportion of Days Attended Scheduled Treatment from Baseline to Post-Intervention at Week 12 | Baseline to Post-Intervention at Week 12.
  Attendance will be defined based on definitions in Petry and colleagues' (2018) and Robinson and colleagues' (2014).
Longest Consecutive Days Attended Scheduled Treatment from Baseline to Post-Intervention at Week 12 | Baseline to Post-Intervention at Week 12.
  Attendance will be defined based on definitions in Petry and colleagues' (2018) and Robinson and colleagues' (2014).
Longest Consecutive Days Absent from Scheduled Treatment from Baseline to Post-Intervention at Week 12 | Baseline to Post-Intervention at Week 12.
  Attendance will be defined based on definitions in Petry and colleagues' (2018) and Robinson and colleagues' (2014).
Mean Number of Days Attended Scheduled Treatment from Baseline to Post-Intervention at Week 12 | Baseline to Post-Intervention at Week 12.
  Attendance will be defined based on definitions in Petry and colleagues' (2018) and Robinson and colleagues' (2014).
Total Number of Days Attended Scheduled Treatment from Baseline to Post-Intervention at Week 12 | Baseline to Post-Intervention at Week 12.
  Attendance will be defined based on definitions in Petry and colleagues' (2018) and Robinson and colleagues' (2014).

OTHER OUTCOMES:
Changes in Quality of Life Measured Using the 26-item World Health Organization (WHO) Quality of Life-BREF (WHOQOL-BREF) | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  The WHOQOL-BREF is a 26-item self-report instrument that measures quality of life across four domains: physical health, psychological health, social relationships, and environment.
Differences in Outcome Measures Between Remote and In-Person Delivery of Contingency Management | Baseline to Post-Intervention Week 12.
  To explore whether the pre-specified outcomes differ between participants who choose to attend their contingency management remotely and participants who choose to attend their contingency management in-person.
Differences in Outcomes Between Participants Seeking Treatment for Methamphetamine Use and Participants Seeking Treatment for Substance Use Issues Other Than Methamphetamine Use | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  To explore whether the pre-specified outcomes differ between participants who are seeking treatment for methamphetamine use and participants seeking treatment for substance use issues other than methamphetamine use.
Differences in Costs Between Contingency Management and Treatment-As-Usual | Baseline to Post-Intervention Week 12.
  To explore differences in the costs of providing contingency management for treatment attendance and treatment-as-usual alone.
Differences in Health Service Use Between Contingency Management and Treatment-As-Usual | Baseline to Post-Intervention Week 12 and from Week 12 to Week 15 (3-Month Follow-Up), Week 18 (6-Month Follow-Up), and Week 24 (12-Month Follow-Up).
  To explore differences in health service use between the experimental group which examines contingency management for treatment attendance and the treatment-as-usual alone group as measured by the number of (a) emergency department visits, (b) visits to urgent care centers, (c) hospitalizations, and (d) enrolments in other treatment services.

CONTACTS AND LOCATIONS:
Overall Officials: David C Hodgins, PhD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Adult Addiction Services in Alberta Health Services, Calgary, Alberta
  - Addiction Services Edmonton in Alberta Health Services, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Impacts of Methamphetamine Abuse in Canada: Hearing Before the House of Comm. Standing Committee on Health, 126 Report, 42nd Parliament, 1st Sess. (Nov. 29, 2018).
- [Background] Dozois DJA, Mikail SF, Alden LE, Bieling PJ, Bourgon G, Clark DA, et al. The CPA presidential task force on evidence-based practice of psychological treatments. Canadian Psychology/Psychologie Canadienne. 2014;55(3):153-160.
- [Background] Sackett DL, Rosenberg WM, Gray JA, Haynes RB, Richardson WS. Evidence based medicine: what it is and what it isn't. BMJ. 1996 Jan 13;312(7023):71-2. doi: 10.1136/bmj.312.7023.71. No abstract available. PMID 8555924
- [Background] Petry NM. Contingency management for substance abuse treatment: a guide for implementing this evidence-based practice. New York: Taylor & Francis Group; 2012.
- [Background] Petry NM, Peirce JM, Stitzer ML, Blaine J, Roll JM, Cohen A, Obert J, Killeen T, Saladin ME, Cowell M, Kirby KC, Sterling R, Royer-Malvestuto C, Hamilton J, Booth RE, Macdonald M, Liebert M, Rader L, Burns R, DiMaria J, Copersino M, Stabile PQ, Kolodner K, Li R. Effect of prize-based incentives on outcomes in stimulant abusers in outpatient psychosocial treatment programs: a national drug abuse treatment clinical trials network study. Arch Gen Psychiatry. 2005 Oct;62(10):1148-56. doi: 10.1001/archpsyc.62.10.1148. PMID 16203960
- [Background] Petry NM, Alessi SM, Rash CJ, Barry D, Carroll KM. A randomized trial of contingency management reinforcing attendance at treatment: Do duration and timing of reinforcement matter? J Consult Clin Psychol. 2018 Oct;86(10):799-809. doi: 10.1037/ccp0000330. PMID 30265039
- [Background] Higgins ST, Budney AJ, Bickel WK, Foerg FE, Donham R, Badger GJ. Incentives improve outcome in outpatient behavioral treatment of cocaine dependence. Arch Gen Psychiatry. 1994 Jul;51(7):568-76. doi: 10.1001/archpsyc.1994.03950070060011. PMID 8031230
- [Background] Roll JM, Chudzynski J, Cameron JM, Howell DN, McPherson S. Duration effects in contingency management treatment of methamphetamine disorders. Addict Behav. 2013 Sep;38(9):2455-62. doi: 10.1016/j.addbeh.2013.03.018. Epub 2013 Apr 3. PMID 23708468
- [Background] Andrade LF, Alessi SM, Petry NM. The impact of contingency management on quality of life among cocaine abusers with and without alcohol dependence. Am J Addict. 2012 Jan-Feb;21(1):47-54. doi: 10.1111/j.1521-0391.2011.00185.x. Epub 2011 Nov 18. PMID 22211346
- [Background] Sindelar J, Elbel B, Petry NM. What do we get for our money? Cost-effectiveness of adding contingency management. Addiction. 2007 Feb;102(2):309-16. doi: 10.1111/j.1360-0443.2006.01689.x. PMID 17222286
- [Background] CRISM-Alberta Health Services. Demographics and service utilization patterns of clients enrolled in specialty addiction treatment for amphetamine use, 2012-2018; Edmonton (Alberta): Canadian Research Initiative in Substance Misuse (CRISM); 2019 Jun. 22 p.
- [Background] Robinson SM, Sobell LC, Sobell MB, Leo GI. Reliability of the Timeline Followback for cocaine, cannabis, and cigarette use. Psychol Addict Behav. 2014 Mar;28(1):154-62. doi: 10.1037/a0030992. Epub 2012 Dec 31. PMID 23276315
- [Background] Sobell LC, Sobell MB. Timeline follow-back: a technique for assessing self-reported alcohol consumption. In Litten RZ, Allen JP (eds). Measuring Alcohol Consumption. Totowa, NJ: Humana Press; 1992:41-72. doi: 10.1007/978-1-4612-0357-5_3
- [Background] Agrawal S, Sobell MB, Sobell LC. The timeline followback: a scientifically and clinically useful tool for assessing substance use. In Belli RB, Stafford FP, Alwin DF (eds). Calendar and Time Diary. Sage Publications Inc; 2009:57-68. doi: 10.4135/9781412990295.d8